CLINICAL TRIAL: NCT00902460
Title: A Phase 1, Randomized, 2-Way Crossover, Multiple Dose, Open Label Study Of The Effect Of CP-690,550 On Midazolam Pharmacokinetics In Healthy Volunteers
Brief Title: CP-690,550 and Midazolam Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A3921059
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Healthy Volunteer
Keywords: drug interactions CYP3A4 CYP3A5 midazolam anti-rheumatic agents
MeSH Terms: interventions — Midazolam; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 (Experimental)
  Interventions: Drug: midazolam; CP-690,550 + midazolam
- Treatment Sequence 2 (Experimental)
  Interventions: Drug: CP-690,550 + midazolam; midazolam

INTERVENTIONS:
Drug: midazolam; CP-690,550 + midazolam — Period 1 : 2 mg midazolam oral syrup alone Period 2: 2 mg midazolam oral syrup plus 30 mg CP-690,550 after 6 days of CP-690,550 at 30 mg BID
  Arms: Treatment Sequence 1
Drug: CP-690,550 + midazolam; midazolam — Period 1: 2 mg midazolam oral syrup plus 30 mg CP-690,550 after 6 days of CP-690,550 at 30 mg BID Period 2: 2 mg midazolam oral syrup alone
  Arms: Treatment Sequence 2

SUMMARY:
CP-690,550 and midazolam are metabolized by similar enzymes in the liver. This study is designed to assess whether co-administration of CP-690,500 and midazolam will effect the metabolism of midazolam in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-child bearing potential) subjects

Exclusion Criteria:

* Clinically significant infections within the past 3 months
* History of previously untreated infection with Mycobacterium tuberculosis
* Positive screening test for hepatitis B surface antigen, anti-hepatitis C antibody, or human immunodeficiency virus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
AUCinf of midazolam | 10 Days

SECONDARY OUTCOMES:
AUClast, Cmax, Tmax, t1/2 of midazolam | 10 Days
Vital signs, laboratory tests and adverse events | 10 Days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921059&StudyName=CP-690%2C550%20and%20Midazolam%20Drug-Drug%20Interaction%20Study